CLINICAL TRIAL: NCT06129942
Title: Light Therapy in Parkinson's Disease: a Prospective, Observational Study
Brief Title: Light Therapy in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chun-Feng Liu, Professor, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JD-LK2020062-R02
Record Dates: First submitted 2021-08-19; First posted 2023-11-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Sleep Disorder; Circadian Rhythm Disorders
MeSH Terms: conditions — Parkinson Disease; Sleep Wake Disorders; Chronobiology Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dim light group (Placebo Comparator): treated with the placebo device which operates with one intensity of 300 lux * 1 month
  Interventions: Device: Dim Light box
- Bright light group (Experimental): treated with the experimental device which operates with one intensity of 10,000 lux * 1 month
  Interventions: Device: Bright light box

INTERVENTIONS:
Device: Bright light box — The light box uses a spectrally transparent prism diffuser, which can block ultraviolet rays, but will not affect the quality of the filtered light and will not turn yellow. The distance between the light box and the patient should not exceed 65cm.PD patients are selected for light intervention of different intensities. The experimental group is treated with 10,000 Lux intensity. The treatment time is 1 hour each day from 08:00-11:00 in the morning and 17:00-19:00 in the afternoon lasting for a month. The patient is asked to move under the light source, but should not fall asleep.
  Arms: Bright light group
Device: Dim Light box — The light box uses a spectrally transparent prism diffuser, which can block ultraviolet rays, but will not affect the quality of the filtered light and will not turn yellow. The distance between the light box and the patient should not exceed 65cm.PD patients are selected for light intervention of different intensities. The control group is treated with 300 Lux intensity. The treatment time is 1 hour each day from 08:00-11:00 in the morning and 17:00-19:00 in the afternoon lasting for a month. The patient is asked to move under the light source, but should not fall asleep.
  Arms: Dim light group

SUMMARY:
The aim of this randomized controlled trial (RCT) is to clarify the effect of bright light therapy on motor symptoms and sleep disorders in patients with Parkinson's disease.

DETAILED DESCRIPTION:
As the most important biologic rhythm timer, exogenous light supplement has certain benefits for the improvement of sleep quality and dementia. At present, it is gradually used in sleep and neuropsychiatric diseases. In an open study, 120 patients with PD received 4000 to 6000 lux of light, for 60 minutes before habitual bedtime. The patients were followed up for several months to 8 years, and it found the patients who persisted in the treatment improved their mood, anxiety and motor function. Clinical studies have confirmed the safety and effectiveness of light in improving insomnia and daytime sleepiness of PD patients. It was found that strong light can significantly improve the patients' motor and non-motor symptoms. However, these findings have not been reported in Chinese PD patients. The aim of this randomized controlled trial (RCT) is to clarify the effect of bright light therapy on motor symptoms and sleep disorders in patients with Parkinson's disease and explore the possible mechanism.

ELIGIBILITY:
Inclusion Criteria:

* According to the criteria of PD diagnosis of the MDS, PD patients were selected as the research object. The clinical symptoms of PD patients were consistent with Hoehn and Yahr stages 2-3.
* All PD patients have maintained stable drug treatment for at least one month, signed clinical informed consent and agreed not to adjust drugs throughout the light test and follow-up period.

Exclusion Criteria:

* Using hypnotic or stimulating drugs.
* Using antidepressants, except stable drugs maintained for more than three months;
* Visual impairment, such as cataract, glaucoma, blindness, etc;
* Cognitive impairment (MMSE < 24);
* There are uncontrollable hallucinations and mental diseases;
* There are sleep phase delay / advance syndrome, shift work, jet lag, etc

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-05-16 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in total sleep time(TST) by polysomnography (PSG) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  Total sleep time is the sum of sleep time in each period. This outcome reflects change of patients' sleep quality.
Changes from baseline in sleep efficient by polysomnography (PSG) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  Sleep efficiency is the ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed. This outcome reflects change of patients' sleep quality.
Change from baseline in REM sleep without atonia by (RWA) polysomnography (PSG) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  REM sleep without atonia (RWA) is the PSG finding of persistent muscle tone during REM sleep, resulting in paroxysmal phasic or tonic EMG activity. Together with dream-enacting behavior (DEB), RSWA is a necessary diagnostic criterion of REM sleep behavior disorder (RBD). This outcome reflects change of RBD severity.
Change from baseline in sleep onset latency polysomnography (PSG) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  Sleep latency is the amount of time it takes patients to go from being fully awake to sleeping. Patients' sleep latency and how quickly they reach rapid eye movement (REM) sleep can be indicators of the amount and quality of sleep they are getting.
Change from baseline in Periodic Limb Movement during Sleep(PLMS) by polysomnography (PSG) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  Periodic limb movement during sleep (PLMS) is is described as a stereotypical involuntary movement during sleep. In particular, presenting more than 15 periodic limb movements per hour is related to daytime sleepiness due to low sleep quality. This outcome reflects change of patients' sleep quality.
Changes from baseline in duration and percentage of each sleep stage by polysomnography (PSG) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  Changes in the length and percentage of N1, N2, N3 and REM sleep,which reflect changes in sleep structure.
Changes from baseline in slow wave activity(SWA) and slow wave energy(SWE) by polysomnography (PSG) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  SWA and SWE are indicators of sleep depth and homeostasis in PSG.

SECONDARY OUTCOMES:
Changes from baseline in MDS Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  MDS Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an effective tool to evaluate the severity of motor symptoms in patients with Parkinson's disease (PD).Each item is simply given a 5- point score: 0 (Absent) to 4 (Marked in amplitude and present most of the time).The higher the MDS-UPDRS score is, the worse the symptoms are.
Changes form baseline in Hoehn-Yahr scale at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  In H-Y scale, PD is divided into 5 stages according to the range and extent of motor symptoms. The higher the H-Y scale is, the worse the symptoms are.
Changes form baseline in PDSS-2 score scale at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  The Parkinson's Disease Sleep Scale-2(PDSS-2) assesses a wide spectrum of disease-specific sleep problems.
Changes form baseline in Pittsburgh sleep quality index (PSQI) score at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  The Pittsburgh sleep quality index (PSQI) is widely used to measure sleep quality. The best cut-off score was 7. The higher the PSQI score is, the worse the sleep quality is.
Changes from baseline in REM sleep behavior disorder questionnaire-Hong Kong (RBDQ-HK) score at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  REM sleep behavior disorder questionnaire-Hong Kong (RBDQ-HK) is widely used to assess the severity of RBD. The higher RBD-HK score is, the worse the symptoms are. In East China, the best cut-off value for RBDQ-HK was located at 17 with a sensitivity of 85% and specificity of 81% (AUC = 0.892) .
Changes from baseline in Epworth sleepiness scale (ESS) score at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  The Epworth sleepiness scale (ESS) measures daytime sleepiness. The best cut-off score was 10.The higher the ESS score is, the worse the excessive sleepiness symptoms are.
Changes from baseline in Morningness-Eveningness Questionnaire (MEQ) score at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  The Morningness-Eveningness Questionnaire (MEQ) is the most widely known questionnaire to assess circadian preference. Cut-off points were evaluated: a range of 14-52 for Evening types, 53-64 for neither types, and 65-86 for Morning types.
Changes from baseline in Hamilton Anxiety Scale(HAMA) score at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  The Hamilton Anxiety Scale(HAMA) is a widely used interview scale to measure the severity of a patient's anxiety . The HAMA score can range from 0 to 56. The higher the HAMA score is, the worse the symptoms are. The best cut-off score was14.
Changes from baseline in Hamilton Depression Scale-24(HAMD-24) score at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  The Hamilton Depression Scale-24(HAMD-24) is a test measuring the severity of depressive symptoms in individuals. The HAMA score can range from 0 to 56. The higher the HAMA score is, the worse the symptoms are.An optimal HAMD-24 cut-off score for distinguishing between patients with and without a depressive disorders was found to be 9/10,with a high area under the curve(AUC) (0.91) indicating excellent discrimination.
Changes in Montreal Cognitive Assessment (MoCA) score at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  Montreal Cognitive Assessment (MoCA) is widely used to assess cognitive dysfunction. The MoCA score can range from 0 to 30.The best cut-off score was 26. The higher the MoCA score is, the better the cognitive function is.
Changes from baseline in Non-Motor Symptoms Questionnaire at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  Non-Motor Symptoms Questionnaire(NMSQ)contains 30 items and requires patients to answer "yes" and "no" according to their own situation in the last month. It is widely used in the assessment of PD patients' non motor symptoms.
Changes from baseline in Parkinson's Disease Questionnaire (PDQ-39) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  The Parkinson's Disease Questionnaire (PDQ-39) is the most frequently used disease-specific health status measure.PDQ-39 total score equal or above 47 was the optimal cut-off associated with a high caregiver strain with a sensitivity of 83% and a specificity of 64% .
Changes from baseline in Fatigue Severity Scale (FSS) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  The Fatigue Severity Scale (FSS) is a scale used in the evaluation of fatigue that affects patients. A list of 9 statements is provided. The best cut-off score was 4.
Changes from baseline in electroencephalogram(EEG) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  Amplitudes of various frequency bands in each cortical region of EEG reflects change of cortical activity.
Changes from baseline in the rhythmic level of melatonin in serum and saliva at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  We collected saliva of participants in sections for 24 hours (6:00, 9:00, 12:00, 15:00, 18:00, 19:00, 20:00, 21:00, 22:00, 23:00, ten time points in total) and serum（8：00，20：00）to detect the level of melatonin. This outcome reflects change of biological rhythm.
Changes from baseline in the rhythmic level of cortisol in serum and saliva at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  We collected saliva of participants in sections for 24 hours (6:00, 9:00, 12:00, 15:00, 18:00, 19:00, 20:00, 21:00, 22:00, 23:00, ten time points in total) and serum（8：00，20：00）to detect the level of cortisol. This outcome reflects change of biological rhythm.
Changes from baseline in functional magnetic resonance(fMRI) at the end of each intervention period | visit1(baseline),visit2(4th week),visit3(8th week),visit4(12th week)
  The functional connections between each brain region and brain network analysis of fMRI reflects change of brain network.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Feng Liu, PhD, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fox SH, Katzenschlager R, Lim SY, Barton B, de Bie RMA, Seppi K, Coelho M, Sampaio C; Movement Disorder Society Evidence-Based Medicine Committee. International Parkinson and movement disorder society evidence-based medicine review: Update on treatments for the motor symptoms of Parkinson's disease. Mov Disord. 2018 Aug;33(8):1248-1266. doi: 10.1002/mds.27372. Epub 2018 Mar 23. PMID 29570866
- [Background] Li Z, Tian T. Light Therapy Promoting Dopamine Release by Stimulating Retina in Parkinson Disease. JAMA Neurol. 2017 Oct 1;74(10):1267-1268. doi: 10.1001/jamaneurol.2017.1906. No abstract available. PMID 28806435
- [Background] Rutten S, Vriend C, Smit JH, Berendse HW, Hoogendoorn AW, van den Heuvel OA, van der Werf YD. A double-blind randomized controlled trial to assess the effect of bright light therapy on depression in patients with Parkinson's disease. BMC Psychiatry. 2016 Oct 21;16(1):355. doi: 10.1186/s12888-016-1050-z. PMID 27769202
- [Background] Paus S, Schmitz-Hubsch T, Wullner U, Vogel A, Klockgether T, Abele M. Bright light therapy in Parkinson's disease: a pilot study. Mov Disord. 2007 Jul 30;22(10):1495-1498. doi: 10.1002/mds.21542. PMID 17516492
- [Background] Riemersma-van der Lek RF, Swaab DF, Twisk J, Hol EM, Hoogendijk WJ, Van Someren EJ. Effect of bright light and melatonin on cognitive and noncognitive function in elderly residents of group care facilities: a randomized controlled trial. JAMA. 2008 Jun 11;299(22):2642-55. doi: 10.1001/jama.299.22.2642. PMID 18544724
- [Background] Rutten S, Vriend C, Smit JH, Berendse HW, van Someren EJW, Hoogendoorn AW, Twisk JWR, van der Werf YD, van den Heuvel OA. Bright light therapy for depression in Parkinson disease: A randomized controlled trial. Neurology. 2019 Mar 12;92(11):e1145-e1156. doi: 10.1212/WNL.0000000000007090. Epub 2019 Feb 15. PMID 30770426
- [Background] Moges H, Vasconcelos OM, Campbell WW, Borke RC, McCoy JA, Kaczmarczyk L, Feng J, Anders JJ. Light therapy and supplementary Riboflavin in the SOD1 transgenic mouse model of familial amyotrophic lateral sclerosis (FALS). Lasers Surg Med. 2009 Jan;41(1):52-9. doi: 10.1002/lsm.20732. PMID 19143012
- [Background] Videnovic A, Klerman EB, Wang W, Marconi A, Kuhta T, Zee PC. Timed Light Therapy for Sleep and Daytime Sleepiness Associated With Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2017 Apr 1;74(4):411-418. doi: 10.1001/jamaneurol.2016.5192. PMID 28241159
- [Result] Muntean ML, Benes H, Sixel-Doring F, Chaudhuri KR, Suzuki K, Hirata K, Zimmermann J, Trenkwalder C. Clinically relevant cut-off values for the Parkinson's Disease Sleep Scale-2 (PDSS-2): a validation study. Sleep Med. 2016 Aug;24:87-92. doi: 10.1016/j.sleep.2016.06.026. Epub 2016 Aug 24. PMID 27810191
- [Result] Opara J, Malecki A, Malecka E, Socha T. Motor assessment in Parkinson;s disease. Ann Agric Environ Med. 2017 Sep 21;24(3):411-415. doi: 10.5604/12321966.1232774. Epub 2017 May 11. PMID 28954481
- [Result] Shen SS, Shen Y, Xiong KP, Chen J, Mao CJ, Huang JY, Li J, Han F, Liu CF. Validation study of REM sleep behavior disorder questionnaire-Hong Kong (RBDQ-HK) in east China. Sleep Med. 2014 Aug;15(8):952-8. doi: 10.1016/j.sleep.2014.03.020. Epub 2014 May 14. PMID 24938584
- [Result] Torbey E, Pachana NA, Dissanayaka NN. Depression rating scales in Parkinson's disease: A critical review updating recent literature. J Affect Disord. 2015 Sep 15;184:216-24. doi: 10.1016/j.jad.2015.05.059. Epub 2015 Jun 10. PMID 26114228
- [Result] Oguh O, Kwasny M, Carter J, Stell B, Simuni T. Caregiver strain in Parkinson's disease: national Parkinson Foundation Quality Initiative study. Parkinsonism Relat Disord. 2013 Nov;19(11):975-9. doi: 10.1016/j.parkreldis.2013.06.015. Epub 2013 Jul 18. PMID 23871587
- [Result] Martinez-Martin P, Rodriguez-Blazquez C, Mario Alvarez, Arakaki T, Arillo VC, Chana P, Fernandez W, Garretto N, Martinez-Castrillo JC, Rodriguez-Violante M, Serrano-Duenas M, Ballesteros D, Rojo-Abuin JM, Chaudhuri KR, Merello M. Parkinson's disease severity levels and MDS-Unified Parkinson's Disease Rating Scale. Parkinsonism Relat Disord. 2015 Jan;21(1):50-4. doi: 10.1016/j.parkreldis.2014.10.026. Epub 2014 Nov 5. PMID 25466406